CLINICAL TRIAL: NCT06746220
Title: Effect of Physical Activity and/or Probiotics on Body Composition and Physiological Parameters in Women
Acronym: AP-Pro-Fem
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHUO-2024-01
Record Dates: First submitted 2024-09-04; First posted 2024-12-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy Women
Keywords: Microbiota; Probiotics; Physical activity; Health; women
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Therapeutics; Probiotics

STUDY DESIGN:
Intervention Model Description: This is a prospective, comparative, double-blind, randomized, monocentric study to explore effects of PA and/or PS on healthy women.
Who Masked: Participant, Investigator
Masking Description: Open label for physical activity or no-physical activity (A versus T groups). Double-blind for placebo/probiotic supplementation (+ versus - groups)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A+ group (probiotic and physical activity) (Experimental): Microbiota sample Salivary sample Quality of life questionnaires Nutritional evaluation Assessment of physical health Physical activity Treatment with placebo or probiotic
  Interventions: Other: Microbiota sample; Other: Salivary sample; Other: Quality of life questionnaires; Other: Nutritional evaluation; Other: Assessment of physical health; Other: Physical activity; Other: Treatment with placebo or probiotic
- A- group (probiotic and non-physical activity) (Experimental): Microbiota sample Salivary sample Quality of life questionnaires Nutritional evaluation Assessment of physical health Physical activity Treatment with placebo or probiotic
  Interventions: Other: Microbiota sample; Other: Salivary sample; Other: Quality of life questionnaires; Other: Nutritional evaluation; Other: Assessment of physical health; Other: Physical activity; Other: Treatment with placebo or probiotic
- T+ group (placebo and physical activity) (Experimental): Microbiota sample Salivary sample Quality of life questionnaires Nutritional evaluation Assessment of physical health Physical activity Treatment with placebo or probiotic
  Interventions: Other: Microbiota sample; Other: Salivary sample; Other: Quality of life questionnaires; Other: Nutritional evaluation; Other: Assessment of physical health; Other: Treatment with placebo or probiotic
- T- group (placebo and non-physical activity) (Experimental): Microbiota sample Salivary sample Quality of life questionnaires Nutritional evaluation Assessment of physical health Physical activity Treatment with placebo or probiotic
  Interventions: Other: Microbiota sample; Other: Salivary sample; Other: Quality of life questionnaires; Other: Nutritional evaluation; Other: Assessment of physical health; Other: Treatment with placebo or probiotic

INTERVENTIONS:
Other: Microbiota sample — Microbiota sample: one sample at inclusion and one sample at the end of the study
Other: Salivary sample — Salivary sample: one sample at inclusion and one sample at the end of the study. In the morning, on an empty stomach.
Other: Quality of life questionnaires — Quality of life questionnaires: 5 auto-questionnaires to be filled at inclusion and at the end of the study
Other: Nutritional evaluation — Nutritional evaluation: food diary completed by participants for 3 consecutive days at inclusion and at the end of the study
Other: Assessment of physical health — Assessment of physical health : 3 tests to assess strength and endurance. These tests will be performed at inclusion and at the end of the study.
Other: Physical activity — Physical activity: 2 sessions per week for 6 weeks. For each session, 45 minutes of physical activity consisting of muscle strengthening and endurance exercises.
  Arms: A+ group (probiotic and physical activity); A- group (probiotic and non-physical activity)
Other: Treatment with placebo or probiotic — Treatment with placebo or probiotic: 1 capsule per day during 42 consecutive days. In the morning, on an empty stomach with a large glass of water 20 minutes before the meal

SUMMARY:
This is a prospective, comparative, double-blind, randomized, monocentric study.

The objective of this project is to evaluate the effects on health of probiotic supplementation (PS) with or without physical activity (PA). Participants who meet the study criteria will be randomized into 4 groups: probiotic and physical activity group (A+), probiotic and non-physical activity group (A-), placebo and physical activity group (T+), placebo and non-physical activity group (T-).

The probiotics used are Lactibiane® Reference provided by Pileje Laboratory. The study population are healthy women (university students) who do not practice sports. A total of 120 participants will participate.

At inclusion, each participant will undergo a medical examination, collect microbiota and salivary samples and perform different tests (questionnaires, assessments of strength and endurance). Then, a follow up phase will last 6 weeks. Each participant will receive a pillbox containing capsules (probiotic or placebo in a double-blind manner). Participants which randomized in the PA groups (A+ and A-) will perform 2 physical activity sessions per week for 6 weeks. At the end of this follow up phase, tests conducting during inclusion will be performed again.

DETAILED DESCRIPTION:
Rationale: Nowadays, the intestinal microbiota is recognized as a significant factor in the health of the host organism. It has an impact on the immune system, the hypothalamo-hypophyseal adrenal axis, the overall state of the individual such as body composition and muscle activity. The intestinal microbiota has also an impact on digestion and associated problems. However, its balance is fragile and can be easily disrupted by a diet rich in proteins or carbohydrates, medications, contraceptive use or lack of physical activity (PA).To restore this balance, subjects may modify their diet, take probiotic supplements (PS) or engage in physical activity. Currently, studies remain limited, particularly regarding effects of physical activity and/or probiotic have never been explored especially in women. The objective of this project is therefore to explore effects of PS and/or PA on the mental and physical health of the holobiont.

Method: Each participant will, during an initial visit, undergo a medical examination (ECG, anthropometric measurements) to ensure there are no contraindications to engaging in physical activity or taking probiotics. Then, we will conduct the first collections of intestinal microbiota and salivary cortisol, initial evaluations of anxiety, depression, and self-esteem (indicators of mental health with questionnaires), as well as assessments of strength and endurance (indicators of physical health), body composition, and nutritional parameters. Following this, participants will be assigned to experimental groups, and we will distribute pillboxes containing capsules (probiotic or placebo in a double-blind manner). Participants in the PA groups (A+ and A-) will perform two 45-minute physical activity sessions per week for 6 weeks, consisting of muscle strengthening and endurance exercises. Participants in the sedentary groups (T+ and T-) will be contacted by phone once a week to ensure proper protocol adherence. At the end of the 6 weeks, we will repeat the tests conducted during the initial visit.

Probiotics: The probiotics used are Lactibiane® Reference, composed of 4 probiotic strains (Bifidobacterium longum LA101, Lactobacillus helveticus LA102, Lactobacillus lactis LA103, Streptococcus thermophilus LA104) dosed at 10 billion per capsule provided by Pileje laboratory. Placebos are also provided by Pileje laboratory.

Statistics: Having no proven hypothesis on the effect of physical activity and/or probiotic supplementation on the population, we started with inclusion of 120 participants in total. This will allow to highlight a moderate effect size (0.25) for the primary endpoint, under the hypothesis of an alpha risk of 0.05, with a power of 80%. and representing 20% lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Being female
2. Age ≥ 18 years old
3. Have a BMI between 18.5 and 30 kg/m2
4. Be registered as a student at the University of Orléans
5. Be non-athletic
6. Have no contraindication to the practice of physical activity
7. All participants must sign informed consent before the start of the study

Exclusion Criteria:

1. Smokers >10 cigarettes per day
2. Having treatment for a pathology at the time of inclusion
3. Taking a probiotic supplement during the last month prior to inclusion
4. Practice physical activity regularly (150 minutes/week of moderate physical activity according to the WHO)
5. Participant under guardianship or curators
6. Pregnant or breastfeeding women
7. Menopausal women
8. Allergy to any excipient known to be present in the probiotic or placebo formulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Effect of physical activity on muscle mass in healthy women | Measure of muscle mass will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Assessment of muscle mass with an impedance meter
Effect of probiotic supplementation on muscle mass in healthy women | Measure of muscle mass will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Assessment of muscle mass with an impedance meter

SECONDARY OUTCOMES:
Effect of physical activity on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for endurance
Effect of physical activity on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for upper limb (grip strength)
Effect of physical activity on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for lower limb (horizontal press test)
Effect of probiotic supplementation on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for upper limb (grip strength)
Effect of probiotic supplementation on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for lower limb (horizontal press test)
Effect of probiotic supplementation on physical condition | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Test for endurance
Effect of physical activity on eating behavior | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Eating behavior: food diary completed by participants for 3 consecutive days. Using specific software (nutrilog), analysis of quantitative energy intake (macronutrients and micronutrients)
Effect of probiotic supplementation on eating behavior | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Eating behavior: food diary completed by participants for 3 consecutive days. Using specific software (nutrilog), analysis of quantitative energy intake (macronutrients and micronutrients)
effect of prebiotics naturally present in food on the composition of the microbiota | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  effect of prebiotics: food diary completed by participants for 3 consecutive days. Using specific software (nutrilog), analysis of the content of foods rich in prebiotics (foods rich in fiber) in the diet.
Effect of physical activity on microbiota | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Microbiota: samples of stool with specific kit (MT0001G Gut Alive). Identify bacterial composition with 16S RNA sequencing
Effect of probiotic supplementation on microbiota | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Microbiota: samples of stool with specific kit (MT0001G Gut Alive). Identify bacterial composition with 16S RNA sequencing
. Effect of physical activity on salivary cortisol | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Salivary cortisol: samples of saliva with specific kit ("salitubes"). Free fraction of cortisol will be analysed by Enzyme-linked immunosorbent assays (ELISA)
. Effect of probiotic supplementation on salivary cortisol | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Salivary cortisol: samples of saliva with specific kit ("salitubes"). Free fraction of cortisol will be analysed by Enzyme-linked immunosorbent assays (ELISA)
. Effect of physical activity on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Quality of life with MOS-SF36 questionnaire
. Effect of physical activity on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Anxiety, depression with HAD questionnaire
. Effect of physical activity on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Self-esteem with ISP-25 questionnaire
. Effect of physical activity on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Effects of dietary supplement with EPCA questionnaire
. Effect of physical activity on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Daily physical activity with IPAQ questionnaire
Effect of probiotic supplementation on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Quality of life with MOS-SF36 questionnaire
Effect of probiotic supplementation on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Anxiety, depression with HAD questionnaire
Effect of probiotic supplementation on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Self-esteem with ISP-25 questionnaire
Effect of probiotic supplementation on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Effects of dietary supplement with EPCA questionnaire
Effect of probiotic supplementation on quality of life | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Daily physical activity with IPAQ questionnaire
Effect of physical activity on fat mass | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Fat mass: assessment of fat mass with an impedance meter
Effect of probiotic supplementation on fat mass | Measure of secondary endpoints will be performed at inclusion and at the end of the study (an average of 2 months after inclusion)
  Fat mass: assessment of fat mass with an impedance meter

CONTACTS AND LOCATIONS:
Overall Officials: Virgile AMIOT, Doctor, Principal Investigator — CHU Orléans
Locations (1):
- Center Hospitalier Universitaire d'Orléans, Orléans, France

REFERENCES:
- [Background] Abenavoli L, Scarpellini E, Colica C, Boccuto L, Salehi B, Sharifi-Rad J, Aiello V, Romano B, De Lorenzo A, Izzo AA, Capasso R. Gut Microbiota and Obesity: A Role for Probiotics. Nutrients. 2019 Nov 7;11(11):2690. doi: 10.3390/nu11112690. PMID 31703257
- [Background] Allen JM, Mailing LJ, Niemiro GM, Moore R, Cook MD, White BA, Holscher HD, Woods JA. Exercise Alters Gut Microbiota Composition and Function in Lean and Obese Humans. Med Sci Sports Exerc. 2018 Apr;50(4):747-757. doi: 10.1249/MSS.0000000000001495. PMID 29166320
- [Background] Alvarez-Arrano V, Martin-Pelaez S. Effects of Probiotics and Synbiotics on Weight Loss in Subjects with Overweight or Obesity: A Systematic Review. Nutrients. 2021 Oct 17;13(10):3627. doi: 10.3390/nu13103627. PMID 34684633
- [Background] Aya V, Florez A, Perez L, Ramirez JD. Association between physical activity and changes in intestinal microbiota composition: A systematic review. PLoS One. 2021 Feb 25;16(2):e0247039. doi: 10.1371/journal.pone.0247039. eCollection 2021. PMID 33630874
- [Background] Aya V, Jimenez P, Munoz E, Ramirez JD. Effects of exercise and physical activity on gut microbiota composition and function in older adults: a systematic review. BMC Geriatr. 2023 Jun 12;23(1):364. doi: 10.1186/s12877-023-04066-y. PMID 37308839
- [Background] Angelakis E, Armougom F, Million M, Raoult D. The relationship between gut microbiota and weight gain in humans. Future Microbiol. 2012 Jan;7(1):91-109. doi: 10.2217/fmb.11.142. PMID 22191449
- [Background] Bastianelli C, Farris M, Bianchi P, Benagiano G. The effect of different contraceptive methods on the vaginal microbiome. Expert Rev Clin Pharmacol. 2021 Jul;14(7):821-836. doi: 10.1080/17512433.2021.1917373. Epub 2021 Apr 23. PMID 33863265
- [Background] Boisseau N, Barnich N, Koechlin-Ramonatxo C. The Nutrition-Microbiota-Physical Activity Triad: An Inspiring New Concept for Health and Sports Performance. Nutrients. 2022 Feb 22;14(5):924. doi: 10.3390/nu14050924. PMID 35267899